CLINICAL TRIAL: NCT01197222
Title: Evaluation of Safety and Efficacy of Using EndoClear-Endoscopic Lens Cleaning Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Oregon Clinic (Other)
Responsible Party: Principal Investigator, Lee Swanstrom, MD, The Oregon Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 940
Record Dates: First submitted 2010-09-08; First posted 2010-09-09 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Laparoscopic Abdominal Surgery
Keywords: Laparoscopic; EndoClear; Lens Cleaning Device

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EndoClear used (Active Comparator): The EndoClear device is used during a laparoscopic abdominal surgery.
  Interventions: Device: EndoClear Lens Cleaning Device
- Control (No Intervention): EndoClear Lens Cleaning Device not used during a laparoscopic abdominal surgery.

INTERVENTIONS:
Device: EndoClear Lens Cleaning Device — EndoClear Lens Cleaning Device is used during a laparoscopic abdominal surgery.
  Other Names: Virtual Ports, Ltd
  Arms: EndoClear used

SUMMARY:
Virtual Ports, Ltd., has developed a lens cleaning device, EndoClear, which is attached to the internal abdominal wall at the beginning of a surgical case and remains in position until completion of the surgery, enabling the surgeon to clean the camera lens without removing it from the abdominal cavity. The purpose of this study is to evaluate the efficacy and safety of using the EndoClear device as a laparoscopic lens cleaning device.

DETAILED DESCRIPTION:
The ability to perform laparoscopic surgery safely and effectively depends on the uninterrupted progression of the operation. Any interruptions to the normal workflow of the procedure threatens to cause distraction which in the least can lengthen the operative time leading to increased hospital operating costs and exposing the patient to unnecessary excess anesthesia and associated risks. At worst, interruptions can cause errors in judgment and/or technique resulting in injury to the patient.

Interruptions in the operating room can take many forms, from conversations to equipment malfunction. The goal of this study is to focus on one particular type of interruption unique to laparoscopic surgery - lens cleaning. It is quite common during the course of the procedure for the laparoscopic scope lens to become obscured by bodily fluids or steam from cautery devices. This necessitates having to remove the camera from the patient, cleaning it outside of the body, applying de-fog solution, reinserting it into the body, and having to reacquire the original camera position and image. This can be quite dangerous particularly in the middle of operative step, such as when there is ongoing bleeding, or when there are sharp or hot instruments within the body. Pilot data from own group demonstrates that the camera may have to be cleaned up to 20 times during a case adding upwards of 10-15 minutes to an operation.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years of age
2. Patients undergoing laparoscopic abdominal surgery

Exclusion Criteria:

1. Patients with known coagulopathy or bleeding tendencies
2. Intra-abdominal abscesses
3. Pregnancy
4. Non-elective laparoscopic surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee L Swanstrom, MD, Principal Investigator — The Oregon Clinic
Locations (1):
- Legacy Good Samaritan, Portland, Oregon, United States